CLINICAL TRIAL: NCT05181501
Title: A Multi-center Clinical Study of Fully Human BCMA Chimeric Antigen Receptor Autologous T (CAR-T) Cell Injection (CT103A) in the Treatment of Newly Diagnosed Subjects With High-risk Multiple Myeloma (FUMANBA-2)
Brief Title: A Study of Fully Human BCMA CAR-T (CT103A) in Patients With Newly Diagnosed High-risk Multiple Myeloma (FUMANBA-2)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT103ACI001
Record Dates: First submitted 2021-11-21; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma
Keywords: newly diagnosed; multiple myeloma; treatment naive; CAR-T
MeSH Terms: conditions — Multiple Myeloma | interventions — CT103A chimeric antigen receptor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CT103A in Newly Diagnosed Subjects With High-risk Multiple Myeloma (Experimental): Fully Human BCMA Chimeric Antigen Receptor Autologous T Cell Injection（CT103A）will be infused at 1.0 x 10^6 CAR+ T cells/kg in newly diagnosed subjects with high-risk multiple myeloma
  Interventions: Drug: Fully human BCMA chimeric antigen receptor autologous T cell injection (CT103A)

INTERVENTIONS:
Drug: Fully human BCMA chimeric antigen receptor autologous T cell injection (CT103A) — CT103A is a customized, BCMA-targeted genetically modified autologous T cell immunotherapy, which can identify and eliminate malignant and normal cells expressing BCMA. CAR specifically recognizes BCMA with single chain fragment variable (ScFv), and promotes the activation, proliferation, cytokine secretion and target cell killing of CAR-T through the CD3ζ domain. And 4-1BB enhances the expansion and persistence of CT103A.
  CT103A will be infused at 1.0×10^6 /kg via intravenous drip within 24h to 72h after chemotherapy conditioning regimen at the recommended infusion rate of 3-5 mL/min.
  Other Names: CT103A

SUMMARY:
This study is a multi-center, single-arm clinical study to evaluate the efficacy, safety, pharmacokinetics and pharmacodynamic characteristics of CT103A as the first-line treatment in newly diagnosed high-risk multiple myeloma subjects with induction chemotherapy as bridging therapy.

DETAILED DESCRIPTION:
Before enrollment, subjects will receive chemotherapy regimen of either Bortezomib-Lenalidomide-Dexamethasone (VRD), Bortezomib-Cyclophosphamide-Dexamethasone (PCD) or Bortezomib-Adriamycin-Dexamethasone (PAD) as induction therapy for 3 cycles. Evaluation will be made after 2 cycles of chemotherapy. If the subject is not intended to have stem cell transplantation or unsuitable for autologous hematopoietic stem cell transplantation (ASCT) as judged by the investigator, he/she will receive the 3rd cycle of chemotherapy. If the subject meets the inclusion criteria, he/she will be enrolled in the study.

Peripheral blood mononuclear cell (PBMC) will be collected to manufacture CT103A. After PBMC collection, the subject will receive another cycle of chemotherapy and evaluated. Lymphodepletion with fludarabine and cyclophosphamide will be performed for three consecutive days. After 1-day rest, subjects will receive a single infusion of CT103A at 1.0 ×10^6 /kg. Subjects will be followed in the study for a minimum of 2 years after CT103A infusion. Long-term follow-up for lentiviral vector safety will be followed for up to 15 years after CT103A infusion.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years old, male or female;
2. Newly diagnosed as high-risk multiple myeloma:

   * Revised Multiple Myeloma International Staging System (R-ISS) stage 3;
   * Double-hit or triple-hit according to FISH test.
3. Presence of measurable lesions during screening according to any of the following criteria:

   * The proportion of primitive naive or monoclonal plasma cells ≥ 5% by bone marrow cytology, bone marrow biopsy histology or flow cytometry;
   * Serum monoclonal protein (M-protein) level: M protein ≥10 g/L for IgG type, M protein ≥5g/L for IgA, IgD, IgM, and IgE type;
   * Urine M protein level ≥200 mg/24 hours;
   * Light chain multiple myeloma without measurable lesions in serum or urine: the affected serum free light chain ≥100 mg/L with abnormal serum κ/λ free light chain ratio;
4. ECOG score of 0 or 1;
5. Expected survival time ≥ 12 weeks;
6. Subjects must have appropriate organ functions and meet all the following laboratory test requirements before enrollment:

   * Hematology: Absolute neutrophil count (ANC) ≥ 1×10^9/L (prior growth factor support is allowed, but supportive treatment within 7 days before laboratory test is not allowed); Absolute lymphocyte count (ALC) )≥0.3×10^9/L; platelets≥75×10^9/L (blood transfusion support within 7 days before laboratory test is not allowed); hemoglobin ≥60 g/L (without red blood cell [RBC] transfusion within 7 days before laboratory test; recombinant human erythropoietin is allowed);
   * Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×upper limit of normal (ULN); serum total bilirubin≤1.5×ULN;
   * Renal function: creatinine clearance calculated according to Cockcroft-Gault formula≥ 40 ml/min.
   * Coagulation function: fibrinogen ≥1.0 g/L; activated partial thromboplastin time≤1.5×ULN, prothrombin time (PT)≤1.5×ULN;
   * Blood oxygen saturation>91%;
   * Left ventricular ejection fraction (LVEF) ≥50%;
7. Subjects and their spouses agree to take effective tools or contraceptive measures (safe period contraception is not included) from the time the subject signs the informed consent form until one year after the CAR-T cell infusion.

Exclusion Criteria:

1. Patient who needs chronic use of immunosuppressive agents;
2. Patient with hypertension that cannot be controlled by medication;
3. Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade III), severe arrhythmia;
4. Unstable systemic diseases judged by the investigator: including but not limited to severe liver, kidney or metabolic diseases that require drug treatment;
5. Patients with malignant tumors other than multiple myeloma within 5 years before screening, excluding fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and those after radical resection Ductal carcinoma in situ of breast;
6. Patient with a history of solid organ transplantation;
7. Patient who is suspected with or with symptoms of central nervous system invasion by plasma cell tumors;
8. Multiple myeloma patients with plasma cell leukemia;
9. Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and detectable hepatitis B virus (HBV) DNA in peripheral blood; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus ( HCV) RNA positive; human immunodeficiency virus (HIV) antibody positive; cytomegalovirus (CMV) DNA test positive; syphilis test positive;
10. Women who are pregnant or breastfeeding;
11. Patient with mental illness or disturbance of consciousness or central nervous system disease;
12. Major surgery history within 2 weeks before entering the study, or scheduled surgery during the study period or within 2 weeks after the study treatment;
13. Other situations considered unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2039-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of Minimal Residual Disease (MRD)-negative subjects | Up to 2 years after CT103A infusion
  The proportion of subjects who achieve MRD-negativity after CT103A infusion.
Median progression-free survival (mPFS) | Up to 2 years after CT103A infusion
  The median time from the date of CT103A infusion to the date of first disease progression or death from any cause.

SECONDARY OUTCOMES:
Best overall response (BOR) | Up to 2 years after CT103A infusion
  The proportion of subjects who achieve stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) after CT103A infusion.
Median survival (mOS) | Up to 2 years after CT103A infusion
  The median time from the date of CT103A infusion to the date of death from any reason.
Event-free survival (EFS) | Up to 2 years after CT103A infusion
  The time from date of CT103A infusion to the date of death from any reason, relapse, treatment failure, disease progression or initiation of other anti-tumor treatment, whichever comes first;
Duration of response (DOR) | Up to 2 years after CT103A infusion
  The time from the first assessment of sCR or CR or VGPR or PR to the first assessment of disease progression or death from any cause;
Safety endpoint | Up to 2 years after CT103A infusion
  Incidence of treatment-emergent adverse events (TEAE) and Treatment-related adverse events (TRAE).
Pharmacokinetic(PK) endpoint | Up to 90 days after CT103A infusion
  The maximum CT103A concentration and the copy number of the lentiviral vector (vector copy number, VCN) in peripheral blood (Cmax)
PK endpoint - Tmax | Up to 90 days after CT103A infusion
  The time to reach the maximum concentration (Tmax)
PK endpoint - AUC 0 to 28d and AUC 0 to 90d | Up to 90 days after CT103A infusion
  The area under the concentration time curve from time zero to day 28 (AUC0-28d) and from time zero to day 90 (AUC0-90d)
Levels of Soluable BCMA | Up to 90 days after CT103A infusion
  The levels of soluble BCMA in peripheral blood at each time point.
PD endpoint | Up to 90 days after CT103A infusion
  The levels of cytokines (IL-6, serum ferritin, etc.) in peripheral blood at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Chen, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Bing Chen, M.D., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (4):
- China (4):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu